CLINICAL TRIAL: NCT05324839
Title: A Multicenter, Prospective, Double-Blinded, Randomized, Parallel-Group, Dose-Ranging Study of Botulinum Toxin Type A Treatment of Wrinkles in Asian
Brief Title: A Study of Botulinum Toxin Type A Treatment of Wrinkles in Asian
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Qing-FengLi Li,MD, professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH9H-2022-T221-2
Record Dates: First submitted 2022-03-09; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Botulinum Toxin, Type A
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- score 1 before injection (Experimental): We injected 1-5 u of BoNTA into score 1 crow's feet lines before being included
  Interventions: Drug: Botulinum toxin type A
- score 2 before injection (Experimental): 2-6 u of BoNTA into score 2 crow's feet lines
  Interventions: Drug: Botulinum toxin type A
- score 3 before injection (Experimental): 3-10 u of BoNTA into score 3 crow's feet lines
  Interventions: Drug: Botulinum toxin type A
- score 4 before injection (Experimental): 5-15 u of BoNTA into score 4 crow's feet lines.
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — injecting different dosage to different group

SUMMARY:
OBJECTIVES： The aim of this randomized, parallel-group, double-blinded controlled multicenter clinical trial is to determine the proper dosage of botulinum toxin type A in Asian, and provide evidence-based proof.

METHODS: 250 patients were included in this study, first, trained observers assessed their wrinkle severity according to the 5-grade Wrinkle Severity Rating Scale before injecting botulinum toxin type A, then we injected different dosages to patients with the different pre-injection scores. All patients were followed up for up to one year. Logistic regression was built, the chi-square test was performed, and R square and p-value are used for evaluation.

DETAILED DESCRIPTION:
This was a self-reported, randomized, parallel-group, double-blinded controlled multicenter clinical trial. It was conducted in Wuhan, Shanghai, and Dongguan, China, at the plastic and reconstructive surgery, and approved by the ethics committee of Shanghai Ninth People's Hospital, affiliated to Shanghai Jiao Tong University School of Medicine. All patients were fully informed about the study in accordance with the applicable regulations and International Conference on Harmonisation Good Clinical Practices guidelines and gave written informed consent before the study. The main inclusion criteria were: 1. Chinese males or females aged over 18 years old who want to accept medical removal of the wrinkle; 2. noticeable symmetrical wrinkles on both sides of the face (grade 1-4 on the 5-grade Wrinkles Severity Rating Scale); 3. female patients must take a pregnancy test to prove they are not pregnant, and they are also asked to use a method of contraception 30 days before inclusion into the group and to use a reliable method of contraception throughout the entire study; 4. patients should not accept other forms of cosmetic intervention and agree to refrain from participation in any other clinical trials that may interrupt the study. The main exclusion criteria were: 1. the wrinkle severity of any site or both sites are either grade 0 or 5 on the 5-grade Wrinkle Severity Rating Scale. 2. the presence of facial hair that may influence the observation of wrinkle severity; 3. the area of injection had an apparent acne scar, active inflammation, infection, cancer or premalignancy, or untreated wound; 4. patients who had facial plastic surgery, tissue transplant, silica gel, liposome (fat) injection, or other permanent or semi-permanent dermal filler; 5. patients who had any type of Botox injection in the last year or were injected more than 3 times.

ELIGIBILITY:
Inclusion Criteria:

* 1. Chinese males or females aged over 18 years old who want to accept medical removal of the wrinkle;
* 2. Noticeable symmetrical wrinkles on both sides of the face (grade 1-4 on the 5-grade Wrinkles Severity Rating Scale);
* 3. Female patients must take a pregnancy test to prove they are not pregnant, and they are also asked to use a method of contraception 30 days before inclusion into the group and to use a reliable method of contraception throughout the entire study;
* 4. Patients should not accept other forms of cosmetic intervention and agree to refrain from participation in any other clinical trials that may interrupt the study.

Exclusion Criteria:

* 1. The wrinkle severity of any site or both sites are either grade 0 or 5 on the 5-grade Wrinkle Severity Rating Scale.
* 2. The presence of facial hair that may influence the observation of wrinkle severity;
* 3. The area of injection had an apparent acne scar, active inflammation, infection, cancer or premalignancy, or untreated wound;
* 4. Patients who had facial plastic surgery, tissue transplant, silica gel, liposome (fat) injection, or other permanent or semipermanent dermal filler;
* 5. Patients who had any type of Botox injection in the last year or were injected more than 3 times.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2014-03-01 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
The change of wrinkle serenity rating scale after 2 weeks | Two weeks after injecting BoNTA
  Compare wrinkle severity according to the 5-grade Wrinkle Severity Rating Scale 2 weeks after Botox injection
The change of wrinkle serenity rating scale after one month | One month after injecting BoNTA
  Compare wrinkle severity according to the 5-grade Wrinkle Severity Rating Scale one month after Botox injection
The change of wrinkle serenity rating scale after three months | Three months after injecting BoNTA
  Compare wrinkle severity according to the 5-grade Wrinkle Severity Rating Scale three months after Botox injection
The change of wrinkle serenity rating scale after six months | Six months after injecting BoNTA
  Compare wrinkle severity according to the 5-grade Wrinkle Severity Rating Scale six months after Botox injection
The change of wrinkle serenity rating scale after nine months | Nine months after injecting BoNTA
  Compare wrinkle severity according to the 5-grade Wrinkle Severity Rating Scale nine months after Botox injection
The change of wrinkle serenity rating scale after one year | One year after injecting BoNTA
  Compare wrinkle severity according to the 5-grade Wrinkle Severity Rating Scale one year after Botox injection

CONTACTS AND LOCATIONS:
Overall Officials: Yun Xie, M.D., Principal Investigator — Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
the status of the participents
Supporting Information: CSR